CLINICAL TRIAL: NCT03469895
Title: Efficacy of BCR Inhibitors in the Treatment of Autoimmune Cytopenias Associated With Chronic Lymphocytic Leukemia (CLL): A Retrospective Analysis of the French Innovative Leukemia Organization (FILO)
Brief Title: Autoimmune Cytopenia and BcR Inhibitors
Acronym: CABRI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: CABRI-IPC 2017-025
Record Dates: First submitted 2018-03-05; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Autoimmune Cytopenia Associated With Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Autoimmune Cytopenias; BCR inhibitors
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- active CLL treated with ibrutinib or idelalisib for CAI: Patient with CLL Active autoimmune cytopenia Initiation of a treatment with ibrutinib or idelalisib for autoimmune cytopenia.
  The progressive nature of contemporary CAI LLC is not a criterion of exclusion.
  Interventions: Drug: ibrutinib ou idelalisib

INTERVENTIONS:
Drug: ibrutinib ou idelalisib — treatment by ibrutinib or idelalisib for autoimmune cytopenia

SUMMARY:
Efficacy of BCR Inhibitors in the Treatment of Autoimmune Cytopenias Associated with Chronic Lymphocytic Leukemia (CLL): A Retrospective Analysis of the French Innovative Leukemia Organization (FILO)

DETAILED DESCRIPTION:
The investigators of the study propose a card of data collection, validated by the scientific council of the group FILO.

The data to be collected are entered on an e-CRF made available to the investigators on a secure site.

The main data collected are as follows

* anonymized demographic data
* Clinical and Biological Data of CLL at Diagnosis
* Previous treatments of LLC and CAI
* clinical and laboratory data at the time of initiation of BCRi treatment
* response to treatment with BCRi
* tolerance to BCRi treatment
* Progression under treatment with BCRi
* Recent news

ELIGIBILITY:
Inclusion Criteria:

* Patient with CLL
* Active autoimmune cytopenia
* Initiation of a treatment with ibrutinib or idelalisib for autoimmune cytopenia.

Exclusion Criteria:

* Other lymphoid hemopathy B
* Absence of documentation of the autoimmunity of cytopenia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with CLL and active autoimmune cytopenia treated with ibrutinib or idelalisib for autoimmune cytopenia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of B-cell receptor inhibitors on autoimmune cytopenia (AIC) | 1 year
  Regarding autoimmune cytopenias, the responses to treatments were defined as such:
  Complete answer
  * hemoglobin level> 120 g/l without transfusion
  * AND platelet count> 100 G/l
  * AND reticulocytes <100 G/l
  * AND normal LDH level Partial answer
  * hemoglobin <120 g/l but with a gain of 2 g/l, without transfusion
  * OR hemoglobin> 120 g/l with reticulocytes> 100 G/l and or high LDH
  * OR hemoglobin> 120 g/l with reticulocytes and / or LDH levels not available
  * AND OR platelet count between 50 and 100 G/l

SECONDARY OUTCOMES:
Efficacy of B-cell receptor inhibitors on the Chronic lymphocytic leukemia (CLL) | 1 year
  Regarding CLL, the responses were defined according to the IWCLL 2008 criteria. Due to the absence of a medullary assessment biopsy, patients presenting the complete clinical and biological response criteria will be considered in a complete clinical response.
Progression Free Survival (PFS) of the autoimmune cytopenia | 1 year
  Progression Free Survival (PFS) of the autoimmune cytopenia
PFS of the Chronic lymphocytic leukemia | 1 year
  PFS of the Chronic lymphocytic leukemia
Event Free Survival (EFS) | 1 year
  Event Free Survival (EFS)
Time to next treatment (TTNT) | 1 year
  Time to next treatment (TTNT)
Toxicity profile | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Overall survival | 1 year
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse Aurran-Schleinitz, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodgson K, Ferrer G, Montserrat E, Moreno C. Chronic lymphocytic leukemia and autoimmunity: a systematic review. Haematologica. 2011 May;96(5):752-61. doi: 10.3324/haematol.2010.036152. Epub 2011 Jan 17. PMID 21242190
- [Background] Dierickx D, Kentos A, Delannoy A. The role of rituximab in adults with warm antibody autoimmune hemolytic anemia. Blood. 2015 May 21;125(21):3223-9. doi: 10.1182/blood-2015-01-588392. Epub 2015 Mar 31. PMID 25827833
- [Background] D'Arena G, Laurenti L, Capalbo S, D'Arco AM, De Filippi R, Marcacci G, Di Renzo N, Storti S, Califano C, Vigliotti ML, Tarnani M, Ferrara F, Pinto A. Rituximab therapy for chronic lymphocytic leukemia-associated autoimmune hemolytic anemia. Am J Hematol. 2006 Aug;81(8):598-602. doi: 10.1002/ajh.20665. PMID 16823816
- [Background] Reynaud Q, Durieu I, Dutertre M, Ledochowski S, Durupt S, Michallet AS, Vital-Durand D, Lega JC. Efficacy and safety of rituximab in auto-immune hemolytic anemia: A meta-analysis of 21 studies. Autoimmun Rev. 2015 Apr;14(4):304-13. doi: 10.1016/j.autrev.2014.11.014. Epub 2014 Dec 9. PMID 25497766
- [Background] Kaufman M, Limaye SA, Driscoll N, Johnson C, Caramanica A, Lebowicz Y, Patel D, Kohn N, Rai K. A combination of rituximab, cyclophosphamide and dexamethasone effectively treats immune cytopenias of chronic lymphocytic leukemia. Leuk Lymphoma. 2009 Jun;50(6):892-9. doi: 10.1080/10428190902887563. PMID 19391041
- [Background] Rossignol J, Michallet AS, Oberic L, Picard M, Garon A, Willekens C, Dulery R, Leleu X, Cazin B, Ysebaert L. Rituximab-cyclophosphamide-dexamethasone combination in the management of autoimmune cytopenias associated with chronic lymphocytic leukemia. Leukemia. 2011 Mar;25(3):473-8. doi: 10.1038/leu.2010.278. Epub 2010 Dec 3. PMID 21127498
- [Background] Quinquenel A, Willekens C, Dupuis J, Royer B, Ysebaert L, De Guibert S, Michallet AS, Feugier P, Guieze R, Levy V, Delmer A. Bendamustine and rituximab combination in the management of chronic lymphocytic leukemia-associated autoimmune hemolytic anemia: a multicentric retrospective study of the French CLL intergroup (GCFLLC/MW and GOELAMS). Am J Hematol. 2015 Mar;90(3):204-7. doi: 10.1002/ajh.23909. Epub 2015 Jan 16. PMID 25428829
- [Background] Maura F, Visco C, Falisi E, Reda G, Fabris S, Agnelli L, Tuana G, Lionetti M, Guercini N, Novella E, Nichele I, Montaldi A, Autore F, Gregorini A, Barcellini W, Callea V, Mauro FR, Laurenti L, Foa R, Neri A, Rodeghiero F, Cortelezzi A. B-cell receptor configuration and adverse cytogenetics are associated with autoimmune hemolytic anemia in chronic lymphocytic leukemia. Am J Hematol. 2013 Jan;88(1):32-6. doi: 10.1002/ajh.23342. Epub 2012 Oct 31. PMID 23115077
- [Background] Byrd JC, Furman RR, Coutre SE, Burger JA, Blum KA, Coleman M, Wierda WG, Jones JA, Zhao W, Heerema NA, Johnson AJ, Shaw Y, Bilotti E, Zhou C, James DF, O'Brien S. Three-year follow-up of treatment-naive and previously treated patients with CLL and SLL receiving single-agent ibrutinib. Blood. 2015 Apr 16;125(16):2497-506. doi: 10.1182/blood-2014-10-606038. Epub 2015 Feb 19. PMID 25700432
- [Background] Byrd JC, Brown JR, O'Brien S, Barrientos JC, Kay NE, Reddy NM, Coutre S, Tam CS, Mulligan SP, Jaeger U, Devereux S, Barr PM, Furman RR, Kipps TJ, Cymbalista F, Pocock C, Thornton P, Caligaris-Cappio F, Robak T, Delgado J, Schuster SJ, Montillo M, Schuh A, de Vos S, Gill D, Bloor A, Dearden C, Moreno C, Jones JJ, Chu AD, Fardis M, McGreivy J, Clow F, James DF, Hillmen P; RESONATE Investigators. Ibrutinib versus ofatumumab in previously treated chronic lymphoid leukemia. N Engl J Med. 2014 Jul 17;371(3):213-23. doi: 10.1056/NEJMoa1400376. Epub 2014 May 31. PMID 24881631
- [Background] Burger JA, Tedeschi A, Barr PM, Robak T, Owen C, Ghia P, Bairey O, Hillmen P, Bartlett NL, Li J, Simpson D, Grosicki S, Devereux S, McCarthy H, Coutre S, Quach H, Gaidano G, Maslyak Z, Stevens DA, Janssens A, Offner F, Mayer J, O'Dwyer M, Hellmann A, Schuh A, Siddiqi T, Polliack A, Tam CS, Suri D, Cheng M, Clow F, Styles L, James DF, Kipps TJ; RESONATE-2 Investigators. Ibrutinib as Initial Therapy for Patients with Chronic Lymphocytic Leukemia. N Engl J Med. 2015 Dec 17;373(25):2425-37. doi: 10.1056/NEJMoa1509388. Epub 2015 Dec 6. PMID 26639149
- [Background] St Bernard R, Hsia CC. Safe utilization of ibrutinib with or without steroids in chronic lymphocytic leukemia patients with autoimmune hemolytic anemia. Ann Hematol. 2015 Dec;94(12):2077-9. doi: 10.1007/s00277-015-2487-8. Epub 2015 Sep 3. No abstract available. PMID 26334319
- [Background] Manda S, Dunbar N, Marx-Wood CR, Danilov AV. Ibrutinib is an effective treatment of autoimmune haemolytic anaemia in chronic lymphocytic leukaemia. Br J Haematol. 2015 Sep;170(5):734-6. doi: 10.1111/bjh.13328. Epub 2015 Feb 25. No abstract available. PMID 25716177
- [Background] Rogers KA, Ruppert AS, Bingman A, Andritsos LA, Awan FT, Blum KA, Flynn JM, Jaglowski SM, Lozanski G, Maddocks KJ, Byrd JC, Woyach JA, Jones JA. Incidence and description of autoimmune cytopenias during treatment with ibrutinib for chronic lymphocytic leukemia. Leukemia. 2016 Feb;30(2):346-50. doi: 10.1038/leu.2015.273. Epub 2015 Oct 7. PMID 26442611
- [Background] Vitale C, Ahn IE, Sivina M, Ferrajoli A, Wierda WG, Estrov Z, Konoplev SN, Jain N, O'Brien S, Farooqui M, Keating MJ, Wiestner A, Burger JA. Autoimmune cytopenias in patients with chronic lymphocytic leukemia treated with ibrutinib. Haematologica. 2016 Jun;101(6):e254-8. doi: 10.3324/haematol.2015.138289. Epub 2016 Mar 24. No abstract available. PMID 27013651
- [Background] Furman RR, Sharman JP, Coutre SE, Cheson BD, Pagel JM, Hillmen P, Barrientos JC, Zelenetz AD, Kipps TJ, Flinn I, Ghia P, Eradat H, Ervin T, Lamanna N, Coiffier B, Pettitt AR, Ma S, Stilgenbauer S, Cramer P, Aiello M, Johnson DM, Miller LL, Li D, Jahn TM, Dansey RD, Hallek M, O'Brien SM. Idelalisib and rituximab in relapsed chronic lymphocytic leukemia. N Engl J Med. 2014 Mar 13;370(11):997-1007. doi: 10.1056/NEJMoa1315226. Epub 2014 Jan 22. PMID 24450857